CLINICAL TRIAL: NCT05606224
Title: The Effects and Mechanisms of Mindfulness Intervention for Emotional Distress: a Multicenter Randomized Controlled Trial
Brief Title: The Effects and Mechanisms of Mindfulness Intervention for Emotional Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Nanjing Brian Hospital (Other); Capital Medical University (Other); Beijing Tiantan Hospital (Other); Foshan Mental Health Center (Unknown)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCRC2021M01
Record Dates: First submitted 2022-10-20; First posted 2022-11-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Emotional Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iMIED+TAU: internet-based mindfulness intervention for emotional distress plus treatment as usual (Experimental): The internet-based self-help version of the Mindfulness Intervention for Emotional Distress (iMIED) program integrates rationales and practices from the UP and MBIs. Formal mindfulness exercises (e.g., body scan, mindful breathing, and mindful stretching) and informal mindfulness practices (e.g., mindful tooth-brushing) were retrieved from MBIs. In addition, iMIED selected several important tasks from the UP, like practicing tolerating uncomfortable feelings by interoceptive exposure practices (e.g., rapid breathing), identifying avoidant behaviors and emotion-driven behaviors and reducing them step by step, identifying common maladaptive automatic thoughts (e.g., overestimating probability and catastrophizing), and using the above strategies in daily life by completing challenging tasks.
  Interventions: Behavioral: internet-based mindfulness intervention for emotional distress
- TAU-only: treatment as usual (No Intervention): In the current study, TAU consisted of all medicinal and psychological treatments received between baseline and follow-up (about five months). Medicinal treatments included receiving Lorazepam, Olanzapine, Paroxetine Hydrochloride, Sertraline, etc. Psychological treatments included receiving cognitive behavior therapy or psychodynamic therapy.

INTERVENTIONS:
Behavioral: internet-based mindfulness intervention for emotional distress — The internet-based self-help version of the Mindfulness Intervention for Emotional Distress (iMIED) program integrates rationales and practices from the UP and MBIs. Formal mindfulness exercises (e.g., body scan, mindful breathing, and mindful stretching) and informal mindfulness practices (e.g., mindful tooth-brushing) were retrieved from MBIs. In addition, iMIED selected several important tasks from the UP, like practicing tolerating uncomfortable feelings by interoceptive exposure practices (e.g., rapid breathing), identifying avoidant behaviors and emotion-driven behaviors and reducing them step by step, identifying common maladaptive automatic thoughts (e.g., overestimating probability and catastrophizing), and using the above strategies in daily life by completing challenging tasks.
  Arms: iMIED+TAU: internet-based mindfulness intervention for emotional distress plus treatment as usual

SUMMARY:
Traditional offline interventions such as MBCT and MBSR have been implemented in treating patients with emotional disorders and obtained significantly improved clinical outcome. However, these offline interventions require the involvement of a therapist expertized in mindfulness and usually charge a high fee, which may not be accessible and cost-effective for lots of patients with psychological disorders. Fortunately, online self-help interventions can compensate for these disadvantages. Our research team has developed a self-help online mindfulness program targeting emotional distress (i.e., MIED), which has been demonstrated to be effective for individuals with emotional distress in a preliminary study. Since patients with emotional disorders usually suffered from emotional distress, the current study will apply this program to these patients, and investigate its auxiliary effects on patients' psychological and physical health.

The primary aim of the current study is to evaluate the effectiveness of MIED for patients with emotional disorders. To do so, we will use a design in which patients who receive online mindfulness training (MIED) except for treatment as usual (TAU) will be compared with patients who receive TAU alone. We expect the intervention to improve patients' psychopathological symptoms reported by the patients and the clinicians or the research team and increase their overall functioning, positive mental health, and physical health compared to TAU. In addition, previous studies have shown that mindfulness interventions improve psychological symptoms through improving cognitive flexibility, distress tolerance, intolerance of uncertainty, and experiential avoidance. Therefore, the secondary aim of the study is to examine the mediating effect of these factors on the relationships between mindfulness practice and improvements in outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* Diagnosis of emotional disorders, including anxiety disorders (e.g., panic disorder, social anxiety disorder, generalized anxiety disorder), and unipolar depression disorders;
* If taking medication, haven't changed for at least 4 weeks before intervention onset, and no change in medicine is expected;
* Voluntary participation in this study and sign an informed consent form.

Exclusion Criteria:

* No access to the internet;
* Inadequate proficiency in Chinese;
* Previous participation in mindfulness-based programs longer than 6 weeks, and/or current practice of meditation more than once per week;
* A history of schizophrenia or schizoaffective disorder, current organic mental disorders, substance abuse disorder, and pervasive developmental disorders;
* Manifesting with any self-injury or suicidal risks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change of mindfulness | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The 20-item Five-Facet Mindfulness Questionnaire-Short Form, self-report, score s range from 20 to 100, higher scores indicate higher levels of mindfulness
Change of other-reported anxiety | at baseline (T0), at post-intervention (T3), and at 3 (T4) months follow-ups
  Hamilton Anxiety Rating Scale, assessed by the clinicians, scores range from 0 to 56, higher scores indicate higher levels of anxiety
Change of other-reported depression | at baseline (T0), at post-intervention (T3), and at 3 (T4) months follow-ups
  Hamilton Depression Rating Scale, assessed by the clinicians, scores range from 0 to 68, higher scores indicate higher levels of depression
Change of self-reported depression | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Beck Depression Inventory-II, self-report, scores range from 0 to 63, higher scores indicate higher levels of depression
Change of self-reported anxiety symptoms | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Beck Anxiety Inventory, self-report, scores range from 0 to 63, higher scores indicate higher levels of anxiety
Change of psychological distress | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  10-item Kessler Psychological Distress Scale, self-report, scores range from 5 to 50, higher scores indicate higher levels of psychological distress
Change of inner peace | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Inner Peace Scale, self-report, scores range from 0 to 28, higher scores indicate higher levels of inner peace
Change of perceived stress | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Chinese Perceived Stress Scales, self-report, scores range from 0 to 28, higher scores indicate higher levels of inner peace
Change of sleep quality | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Pittsburgh Sleep Quality Index, self-report, scores range from 0 to 21, higher scores indicate worse sleep quality
Change of Depression Severity and Impairment | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Overall Depression Severity and Impairment Scale, self-report, scores range from 0 to 20, higher scores indicate higher levels of depression severity and impairment
Change of Anxiety Severity and Impairment | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Overall Anxiety Severity and Impairment Scale, self-report, scores range from 0 to 20, higher scores indicate higher levels of anxiety severity and impairment
Change of somatic symptoms | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Patient Health Questionnaire-15, self-report, scores range from 0 to 30 higher scores indicate higher levels of somatic symptoms
Change of distress tolerance | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Chinese version of the Distress Tolerance Scale, self-report, scores range from 15 to 75 higher scores indicate higher levels of distress tolerance
Change of Intolerance of Uncertainty | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Intolerance of Uncertainty -Short form, self-report, scores range from 12 to 60, higher scores indicate higher levels of intolerance of uncertainty
Change of experiential avoidance | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Brief Experience Avoidance Questionnaire, self-report, scores range from 15 to 75 higher scores indicate higher levels of experiential avoidance
Change of attention control | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Attention Control Scale, self-report, scores range from 16 to 64 higher scores indicate higher levels of attention control
Change of Cognitive Flexibility | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Cognitive Flexibility Inventory, self-report, scores range from 20 to 100, higher scores indicate higher levels of cognitive flexibility
Change of discomfort intolerance | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Discomfort intolerance Scale, self-report, scores range from 0 to 25 higher scores indicate higher levels of discomfort intolerance

SECONDARY OUTCOMES:
Change of distress tolerance (behavioral indicator1) | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Paced Auditory Serial Addition Task-Computerized, task persistence as the behavioral indicator of emotional distress
Change of distress tolerance (behavioral indicator2) | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Emotional Image Tolerance Task, distress persistence as the behavioral indicator of emotional distress (after selecting "quit," the average time participants viewed the slide before moving on to the next slide)
Change of distress tolerance (behavioral indicator3) | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Mirror tracing task, task persistence as the behavioral indicator of emotional distress

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (4):
- China (4):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Fosha Mental Health Center, Foshan, Guangdong
  - Nanjing Brain Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No